CLINICAL TRIAL: NCT00243698
Title: A Pilot Study Evaluation of the Efficacy of SonoVue to Detect and Characterise Breast Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT03-FT/SEN
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Breast Tumors
Keywords: Contrast-enhanced Ultrasound Sonography; Ultrasound Contrast agents, microbubbles; Breast tumors
MeSH Terms: conditions — Breast Neoplasms | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SonoVue (sulphur hexafluoride microbubbles) — One contrast enhanced ultrasonography using sonovue / 4.8 ml per injection (maximum of 3 injections)

SUMMARY:
Ultrasound is a well-established imaging modality for the evaluation of breast disease.

The investigators' objective is to characterise the properties of an intravascular ultrasonographic contrast agent SonoVue (sulphur hexafluoride microbubbles) to improve the diagnostic value of the ultrasound examination in patients with different breast lesions.

The final purpose of this ultrasonography is to allow the early detection of tumors and to improve the differentiation between benign and malignant lesions.

SonoVue® (sulphur hexafluoride microbubbles) is a microbubbles preparation that is stable, resistant to pressure, and specifically designed to be used as a contrast agent for ultrasound imaging.

Contrast-enhanced ultrasound could provide a non-invasive technique to evaluate the morphology of breast tumour vascularity.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the efficacy of SonoVue® to detect breast lesions and define specific microcirculation patterns in patients with four different type of breast lesions (enlarging fibroadenoma, suspect malignant nodules, microcalcification and large malignant nodules) in comparison with pathological specimens in terms of histology diagnosis and microvessel density evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Woman presenting with: enlarging fibroadenoma (less than 2 cm in diameter or woman over 40 years old with fibroadenoma less than 2 cm in diameter) or suspect malignant nodule (less than 2 cm in diameter) or a cluster of microcalcification or a malignant nodule (size greater than 3 cm) diagnosed with mammography and/or MRI and/or United States (US) examination performed within 1 month before the study.
* Woman scheduled for biopsy or surgery within 1 month from the examination.

Exclusion Criteria:

* Patients who have already performed a biopsy on the lesion during investigation
* Any contraindication to perform a contrast-enhanced MRI examination for the patients presenting with a malignant nodule (size greater than 3 cm)
* Patients previously entered in this study or having received an investigational drug within 30 days prior to admission to this study
* Patients with any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data or of achieving the study objectives (drug dependence, psychiatric disorders, dementia or other reasons)
* Pregnant or nursing female
* Patient known to have a coronary syndrome
* Unstable angina and myocardial infarction
* Acute cardiac failure, Class III/IV cardiac failure
* Severe rhythm disorders
* Acute endocarditis
* Prosthetic valves

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
From contrast-enhanced ultrasound: Time-intensity curves obtained with SonoVue will help the investigators in differentiation of lesions based on different enhancements. | Inclusion period

SECONDARY OUTCOMES:
Histology assessments: Microvessel density assessments to evaluate the total amount of microcirculation and the neoangiogenesis microcirculation present in the samples | inclusion period
Off-line time-intensity curves from contrast-enhanced magnetic resonance imaging (MRI) images (malignant nodule greater than 3 cm in diameter only) | inclusion period

CONTACTS AND LOCATIONS:
Overall Officials: François Tranquart, PR, Study Director — Centre d'Innovation Technologique CHRU Tours; Catherine LABBE, MD, Principal Investigator — CRLCC René Gauducheau 44805 ST HERBLAIN
Locations (1):
- University Hospital of Tours, Tours, France

REFERENCES:
- [Background] Kettenbach J, Helbich TH, Huber S, Zuna I, Dock W. Computer-assisted quantitative assessment of power Doppler US: effects of microbubble contrast agent in the differentiation of breast tumors. Eur J Radiol. 2005 Feb;53(2):238-44. doi: 10.1016/j.ejrad.2004.04.017. PMID 15664287
- [Background] Singh S, Pradhan S, Shukla RC, Ansari MA, Kumar A. Color Doppler ultrasound as an objective assessment tool for chemotherapeutic response in advanced breast cancer. Breast Cancer. 2005;12(1):45-51. doi: 10.2325/jbcs.12.45. PMID 15657523
- [Background] Watermann D, Madjar H, Sauerbrei W, Hirt V, Prompeler H, Stickeler E. Assessment of breast cancer vascularisation by Doppler ultrasound as a prognostic factor of survival. Oncol Rep. 2004 Apr;11(4):905-10. PMID 15010893
- [Background] Martinez AM, Medina CJ, Bustos C, Hernandez JA. Assessment of breast lesions using Doppler with contrast agents. Eur J Gynaecol Oncol. 2003;24(6):527-30. PMID 14658595
- [Result] Cosgrove DO, Kedar RP, Bamber JC, al-Murrani B, Davey JB, Fisher C, McKinna JA, Svensson WE, Tohno E, Vagios E, et al. Breast diseases: color Doppler US in differential diagnosis. Radiology. 1993 Oct;189(1):99-104. doi: 10.1148/radiology.189.1.8372225.